CLINICAL TRIAL: NCT07125014
Title: Frequency and Risk Factors of Post-ERCP Pancreatitis: A Single-Center Experience From South Asia
Brief Title: Frequency and Predictors of Post-ERCP Pancreatitis in a South Asian Tertiary Care Center
Status: Completed | Type: Observational
Sponsor: Nangarhar University (Other)
Responsible Party: Principal Investigator, Rafiullah Hotak, Doctor, Nangarhar University
Other Study IDs: Ref: No.1027/LRH/MTI
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Post-ERCP Pancreatitis
Keywords: Endoscopic retrograde cholangiopancreatography; ERCP complications; Pancreatitis risk factors
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Observational study — This is an observational study with no experimental or therapeutic interventions administered to participants. All data were collected retrospectively from existing hospital records for patients who underwent ERCP between January 2023 and December 2023 at Lady Reading Hospital, Peshawar. No drugs, devices, or procedures were assigned to participants as part of this research.

SUMMARY:
This study was conducted at the Department of Gastroenterology, Lady Reading Hospital, Peshawar, Pakistan, from January 2023 to December 2023. It aimed to determine how often patients develop pancreatitis (inflammation of the pancreas) after undergoing a procedure called endoscopic retrograde cholangiopancreatography (ERCP), and to identify the main factors that increase this risk. We reviewed the medical records of 300 adult patients who had ERCP for various conditions, such as bile duct stones, tumors, and strictures. We assessed patient characteristics, procedure details, and laboratory results to see which factors were linked to post-ERCP pancreatitis. The study found that prolonged cannulation time, injection of contrast into the pancreatic duct, and high levels of C-reactive protein before the procedure were the strongest predictors of this complication. These findings may help doctors identify high-risk patients and take preventive steps to reduce the chances of pancreatitis after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Known chronic pancreatitis
* Pancreatic malignancy
* Pre-existing acute pancreatitis
* Incomplete procedural or laboratory records

Exclusion Criteria:

* Known chronic pancreatitis
* Pancreatic malignancy
* Pre-existing acute pancreatitis
* Incomplete procedural or laboratory records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing ERCP at the Department of Gastroenterology, Lady Reading Hospital, Peshawar, between January 2023 and December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Post-ERCP Pancreatitis | Within 24 hours after ERCP and during hospitalization
  The number and proportion of patients developing post-ERCP pancreatitis (PEP), defined as new or worsened abdominal pain with serum amylase or lipase levels ≥3 times the upper limit of normal within 24 hours after ERCP, requiring hospitalization or prolongation of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- LRH/MTI, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No